CLINICAL TRIAL: NCT01994902
Title: Investigation of Newly Developed 1-and 2-piece Convex Ostomy Products in Subjects With Ileostomy.
Brief Title: Investigation of Newly Developed Ostomy Products in Subjects With Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP232
Record Dates: First submitted 2013-10-18; First posted 2013-11-26 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-12

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Coloplast test product (Experimental): The subjects test:
  test period 1: Coloplast test product test period 2: SenSura Convex Light
  Interventions: Device: Coloplast test product; Device: SenSura Convex Light
- First SenSura Convex Light (Experimental): The subjects test:
  test period 1: SenSura Convex Light test period 2: Coloplast test product
  Interventions: Device: Coloplast test product; Device: SenSura Convex Light

INTERVENTIONS:
Device: Coloplast test product — The Coloplast test product is a newly developed ostomy appliance
Device: SenSura Convex Light — The comparator product is SenSura Convex Light, which is CE-marked and commercially available.
  Other Names: SenSura

SUMMARY:
The aim of the investigation was to investigate the performance and safety of a new ostomy product.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years of age and have full legal capacity.
2. Has had an ileostomy for at least 3 months.
3. Has used a convex ostomy product for the last month.
4. Has given signed informed consent.
5. Has experienced seeping under the baseplate at least three times during the last two weeks.
6. Currently using a SenSura Convex product with midi, maxi or magnum bags.
7. Currently using a 1-piece product or a 2-piece product with a mechanical coupling ("click coupling").
8. Has an ileostomy with a diameter of max 33 mm (1-piece product) or less. Or Has an ileostomy with a diameter of 30 mm (2-piece product) or less.

Exclusion Criteria:

1. Has a loop-ostomy (double-barrel ostomy or ostomy with two outlets).
2. Are pregnant or breastfeeding.
3. Currently receiving, or has within the past 2 months received radio- and/or chemotherapy.
4. Currently receiving, or has within the past month received steroid treatment (adrenocortical hormone) systemically or locally in the peristomal area.
5. Currently suffering from peristomal skin problems i.e. bleeding or broken (weeping) skin.
6. Are currently participating in another clinical intervention study or have previously participated in this one.
7. Has a fistula in the peristomal area or less than 2 cm from the edge of the baseplate.
8. Has known hypersensitivity toward the test product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Carter, Study Director — Coloplast A/S
Locations (29):
- TFS, Søborg, Denmark
- France (8):
  - Hopital du bocage, Dijon
  - Hopital Robert Boulin, Libourne
  - Hopital Claude Huriez, Lille
  - Hopital Nord, Marseille
  - Hopital Cochin, Paris
  - Hopital Tenon, Paris
  - Hopital de Haut Levêque, Pessac
  - CHRU La Milétrie, Poitiers
- Germany (12):
  - BB medica medizinisches, Aachen
  - Sanitätshause reinhold hilscher e.K., Augsburg
  - Patientenberatung Strack e.K., Bad Staffelstein
  - Pro-samed Santitätshaus, Berlin
  - SIEWA coloplast Homecare, Burgdorf, Hanover
  - SIEWA Coloplast Homecare, Freising
  - SIEWA Coloplast homecare, Leinfelden-Echterdingen
  - Schürmaier GmbH &Co, Leipzig
  - Sanitätshaus Fürst GmbH, Passau
  - SIEWA Coloplast Homecare, Saulgrub
  - Sanitäts- und gesundheitshaus Carqueville GmbH, Töppeln
  - Alippi GmbH, Zwickau
- Sykpleierklinikken, Larvik, Norway
- United Kingdom (7):
  - Pilgrim Hospital, Boston
  - Addenbrookes, Cambridge
  - Cheltenham General Hospital, Gloucestershire
  - Lincon Country hospital, Lincoln
  - Charing Cross Hospital, London
  - Kettering General hospital, Northamptonshire
  - west Suffolk Hospital, Suffolk

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 129 subjects were randomized, but two of these subjects were not exposed to a product: one subject had a stoma diameter of 42 mm (violation to inclusion criteria no.8) and one subject had chemotherapy planned (exclusion criteria no.3). 127 subjects were therefore included in the ITT population.
Groups:
- First Coloplast Test Product; Then SenSura Convex Light: The subjects test:
  test period 1: Coloplast test product test period 2: SenSura Convex Light
  .
- First SenSura Convex Light; Then Coloplast Test Product: The subjects test:
  test period 1: SenSura Convex Light test period 2: Coloplast test product
Period: Test Period 1
Arm/Group | First Coloplast Test Product; Then SenSura Convex Light | First SenSura Convex Light; Then Coloplast Test Product
Started | 63 | 64 (Randomisation mistake:a subject randomised to SenSura Convex Light but tested Coloplast test product)
Completed | 57 | 61 (The subject testing Coloplast test product discontinued due to device deficiency with adverse event)
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — device deficiency with adverse event | 0 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — bag too small | 1 | 0
Period: Test Period 2
Arm/Group | First Coloplast Test Product; Then SenSura Convex Light | First SenSura Convex Light; Then Coloplast Test Product
Started | 57 | 61
Completed | 57 | 55
Not Completed | 0 | 6
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Population: Only subjects in the intention to treat population are included in the baseline population. These were the only subjects who tested the products.
Groups:
- Overall Study: The investigation is a cross-over investigation therefore the baseline data is given for the overall study population
Arm/Group | Overall Study
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (14.1)
Gender [Number; unit: participants] — one gender registration was missing
  participants
    Female | 77
    Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The degree of leakage is measured using a 33-point scale measuring leakage under the baseplate, where 0 points represents the best possible outcome (no leakage) and 33 points the worst possible outcome (leakage on the whole baseplate).
Time Frame: 28 +/- 3 days
Population: The results presented above are the intention-to-treat results that were analysed as randomised. However, the adverse events are reported as treated and as 4 subjects did not follow the randomisation order there is a slight discrepancy between the participants number in the outcome and adverse events section.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: baseplates
Groups:
- Coloplast Test Product: Leakage results obtained while subjects tested the Coloplast test product
- SenSura Convex Light: The leakage results obtained while subjects were testing SenSura Convex Light
Arm/Group | Coloplast Test Product | SenSura Convex Light
Number analyzed (Participants) | 124 | 121
Number analyzed (baseplates) | 1967 | 1988
units on a scale | 5.1 (5.8) | 5.8 (5.8)

ADVERSE EVENTS:
Groups:
- Coloplast Test Product: Adverse events reported by subjects testing Coloplast test product
- SenSura Convex Light: Adverse events reported by subjects testing SenSura Convex Light
Arm/Group | Coloplast Test Product | SenSura Convex Light
Serious Adverse Events (participants affected / at risk) | 6/125 | 3/120
Other Adverse Events (participants affected / at risk) | 28/125 | 14/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product (N=125) | SenSura Convex Light (N=120)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) — unlikely related to the device
acute abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — unlikely related to the device
gastrientitis (Infections and infestations) | 1 (1) | 0 (0) — not related to product
stoma operation (revision of stome) (Gastrointestinal disorders) | 1 (1) | 0 (0) — not related to product
obstruction of stoma (Gastrointestinal disorders) | 1 (1) | 0 (0) — not related to product
Blocked stoma (Gastrointestinal disorders) | 0 (0) | 1 (1) — not related to product
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — not related to product
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) — not related to product
Severe sepsis in contex of intra abdominal infection (Infections and infestations) | 0 (0) | 1 (1) — not related to product
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product (N=125) | SenSura Convex Light (N=120)
Skin irritations (Skin and subcutaneous tissue disorders) | 28 (51) | 14 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less